CLINICAL TRIAL: NCT01366131
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of MEGF0444A in Combination With Carboplatin , Paclitaxel and Bevacizumab in Patients With Advanced or Recurrent Non-Squamous Non-Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy for Advanced Disease
Brief Title: Study Evaluating the Safety and Efficacy of MEGF0444A in Combination With Carboplatin, Paclitaxel and Bevacizumab in Patients With Advanced or Recurrent Non-Squamous Non-Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy for Advanced Disease (NILE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEF4984g; GO27811 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — parsatuzumab; Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: MEGF0444A; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- B (Experimental)
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: MEGF0444A — Intravenous repeating dose
  Arms: A
Drug: bevacizumab — Intravenous repeating dose
Drug: carboplatin — Intravenous repeating dose
Drug: paclitaxel — Intravenous repeating dose
Drug: placebo — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of MEGF0444A combined with paclitaxel + carboplatin + bevacizumab therapy in patients with histologically or cytologically documented inoperable, locally advanced, metastatic (Stage IV), or recurrent non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented inoperable (Stage IV) or recurrent non-squamous non-small cell lung cancer (NSCLC). Diagnoses of non-squamous NSCLC that are based on sputum cytology alone are not acceptable. Mixed tumors should be categorized according to the predominant cell type.
* ECOG performance status of 0 or 1
* Life expectancy >12 weeks
* Measurable disease, as defined by RECIST 1.1
* Adequate hematologic and end organ function

Exclusion Criteria:

* Prior therapy (including chemotherapy, antibody therapy, tyrosine kinase inhibitors,radiotherapy, immunotherapy, hormonal therapy or investigational therapy) before Day 1 of Cycle 1 for the treatment of Stage IV or recurrent NSCLC. Patients who received prior adjuvant chemotherapy or radiotherapy for NSCLC are not excluded if the time interval from completion of adjuvant therapy until disease progression is > 12 months.
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent
* Pregnant and lactating women
* Active infection requiring IV antibiotics

Bevacizumab-Specific Exclusions:

* Histologically or cytologically documented inoperable, locally advanced, mixed non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Evidence of tumor invading major blood vessels on imaging
* Evidence of central nervous system (CNS) metastases
* History of stroke or transient ischemic attacks (TIAs) within 6 months prior to Day 1
* Significant vascular disease within 6 months prior to Day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (defined as the time from randomization to the first occurrence of progression based on RECIST 1.1 criteria or death from any cause on study) | Up to 24 months

SECONDARY OUTCOMES:
Objective response (partial response plus complete response) as determined by the Investigator using RECIST 1.1 | Up to 24 months
Duration of objective response (defined as the first occurrence of a documented objective response until the time of progression or death from any cause on study) | Up to 24 months
Overall survival (defined as the time from randomization until death from any cause) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ina Rhee, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (40):
- United States (20):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Santa Monica, California
  - Orlando, Florida
  - Port Saint Lucie, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Burnsville, Minnesota
  - Las Vegas, Nevada
  - Albany, New York
  - Columbus, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Vancouver, Washington
- Australia (3):
  - St Leonards, New South Wales
  - Herston, Queensland
  - Woodville South, South Australia
- Czechia (2):
  - Brno
  - Ostrava - Poruba
- France (6):
  - Le Mans
  - Lyon
  - Marseille
  - Paris
  - Saint-Herblain
  - Toulouse
- Germany (4):
  - Essen
  - Gauting
  - Großhansdorf
  - Halle
- Hungary (3):
  - Budapest
  - Székesfehérvár
  - Tatabánya
- Poland (2):
  - Bydgoszcz
  - Gdansk

REFERENCES:
- [Derived] von Pawel J, Spigel DR, Ervin T, Losonczy G, Barlesi F, Juhasz E, Anderson M, McCall B, Wakshull E, Hegde P, Ye W, Chen D, Chang I, Rhee I, Reck M. Randomized Phase II Trial of Parsatuzumab (Anti-EGFL7) or Placebo in Combination with Carboplatin, Paclitaxel, and Bevacizumab for First-Line Nonsquamous Non-Small Cell Lung Cancer. Oncologist. 2018 Jun;23(6):654-e58. doi: 10.1634/theoncologist.2017-0690. Epub 2018 Feb 7. PMID 29438092